CLINICAL TRIAL: NCT02434900
Title: Vitamin D and Angiogenic Markers in Odense Child Cohort 1: A Prospective Cohort Study on Their Role in Early Pregnancy Adverse Outcome
Brief Title: Vitamin D and Angiogenic Markers in Odense Child Cohort 1
Acronym: VITAM
Status: Active, not recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Christesen, MD, PhD, Associate Professor, Odense University Hospital
Other Study IDs: VITAM1
Record Dates: First submitted 2014-11-20; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Abortion, Spontaneous
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Vitamin D and Angiogenic Marker Study 1:

Vitamin D and angiogenic markers in early pregnancy. Epidemiology and associations to early-pregnancy miscarriage

DETAILED DESCRIPTION:
Overall: The Odense Child Cohort Study (OCC) is a population-based cohort study, comprising pregnant women recruited between January 1st 2010 and December 31st 2012. All women who were pregnant in the municipality of Odense during this time were eligible for participation, and 6,707 women were approached directly with recruitment material.

The study complied with the Helsinki declaration and was approved by the Regional Scientific Ethical Committee for Southern Denmark, no. S-20090130. All participants gave informed consent. From a population base of 6,707 pregnant women, 2,874 (42.9%) enrolled in the OCC up to December 31st, 2012. The children will be followed until 18 years of age.

Serum samples were taken in early pregnancy (GA 2-25 weeks), late pregnancy (GA 26-30 weeks), maternal serum and cord blood at birth, and from the children along with general examinations at ages 3 months, 1 year, 3 years.

Questionnaires were completed by the families in early pregnancy, late pregnancy, after birth, and at the times of clinical examination of the children.

Register data on health variables were further available from the Danish registries.

Objective: The Vitamin D and Angiogenic Marker Study 1 examines the relationship between serum biomarkers 25(OH)D and soluble Fms-like kinase 1 (sFlt-1) and placental growth factor (PlGF) in pregnancy and risk of miscarriage as an adverse outcome in early pregnancy.

Method:

* 25(OH)D analysis: Serum was stored at -80º Celsius until analysis, which was performed by liquid chromatography mass spectrometry (LC-MS/MS). Triple deuterium marked 25(OH)vitamin D3 was added to serum samples as internal standard and deproteinized with ZnSO4 in methanol, centrifuged at 2750 g for 10 minutes, and 100 μl was injected on the TurboFlow column (Thermo Scientific) on the LC-MS/MS. The LC-MS/MS consisted of a Thermo Scientific TLX1 system connected to a Thermo Scientific Vantage TSQ. 25(OH)D2 and 25(OH)D3 were concentrated on a Thermo Scientific Cyclone P 50 x 1.0 mm column and back-flushed on the analytical column, Phenomenex Gemini C18 50 x 3.0 mm and eluted from the analytical column by a gradient. Mobile phases were A: 10 mM NH4Ac in water and B: 10 mM NH4Ac in methanol. Human serum was spiked with appropriate amounts of 25(OH)D2 and 25(OH)D3 in order to produce six point calibration curves (weighed 1/x2) and 3 levels of QC samples (low, mid, high). The method was calibrated against NIST standard 972.25 The C3 epimer of D3 was detected along with D3 and the two were not distinguishable from one another. Lowest detectable concentrations were 0.15 nM for both D2 and D3. Values of D2 and D3 were only considered if above 6.5 nM.
* Measurements for BRAHMS sFlt-1 and PIGF KRYPTOR assays were performed on the fully automated KRYPTOR compact Plus system (KRYPTOR PlGF and KRYPTOR sFlt-1; Thermo Fisher Scientific) according to the manufacturer's instructions. The BRAHMS sFlt-1 and PlGF KRYPTOR assays are homogeneous sandwich immunoassays based on the Trace technology24. The total duration of the assays are 9 minutes (sFlt-1) and 29 minutes (PlGF) and the sample volume is 9 µl, and 70 μl, respectively. The assays are calibrated with recombinant human sFlt-1 and PIGF and standardized against the Quantikine PIGF ELISA (R&D Systems Europe Ltd, Abingdon, UK) and against the sFlt-1 Elecsys assay (Elecsys, Penzberg, Germany). According to the manufacturer's instructions for use, the KRYPTOR sFlt-1 assay covered a measuring range of 22-90,000 pg/ml. The limit of detection is 22 pg/ml and the limit of quantization (functional sensitivity) is 29 pg/ml. The intra- and inter-assay variations at an sFlt-1 concentration of 1540 pg/ml are 0.3% and 0.8%, respectively; at 2988 pg/ml 0.5% and 1.1%; and at 9666 pg/ml 0.5% and 1.0%, respectively. The KRYPTOR PlGF assay covers a measuring range of 3.6-7.000 pg/ml. The limit of detection is 3.6 pg/ml and the limit of quantitation is 6.9 pg/ml. The intra- and inter-assay variations at a PlGF concentration of 35 pg/ml are 4.6% and 7.3%, respectively; at 103 pg/ml 2.1% and 3.1%, and at 430 pg/ml 0.9% and 2.3%, respectively.
* Measurements for Elecsys sFlt-1 and PIGF assays were performed on the fully automated Elecsys system (Elecsys, Penzberg, Germany) according to the manufacturer's instructions. The Elecsys assays are sandwich immunoassays based on the electrochemiluminescence technology. The total duration of the assays is 18 minutes and the sample volume is 20 µl for sFlt-1 and 50 µl for PIGF. The assays are calibrated with recombinant human PIGF and sFlt-1 and standardized against the Quantikine PIGF and vascular endothelial growth factor-R1 ELISAs (R&D Systems, Minneapolis, MN). According to the manufacturer's instructions for use, the Elecsys sFlt-1 assay covers a measuring range from 10-85,000 pg/ml, the Elecsys PIGF assay from 3-10,000 pg/ml. The limit of detection is 10 pg/ml (sFlt-1) and 3 pg/ml (PIGF). The limit of quantization is 15 pg/ml for sFlt-1 and 10 pg/ml for PIGF.

The Vitamin D and Angiogenic Marker Study 1:

Vitamin D and angiogenic markers in early pregnancy. Epidemiology and associations to early-pregnancy miscarriage

* In 1728 serum samples collected in early pregnancy, the levels of serum 25(OH)D were investigated by LC-MS/MS and levels of sFlt-1 and PlGF were determined by immunoassays in 1720 samples. Questionnaire and medical file information was used to determine the factors which were influential on 25(OH)D levels and sFlt/PlGF in early pregnancy by multiple linear regression and logistic regression.
* In 1675 serum samples collected before gestational age 22+0 weeks, analysis was performed to evaluate the predictive properties of sFlt-1 and PlGF levels as biomarkers of miscarriage (n=59).
* In 1684 serum samples collected before gestational age 22+0 weeks, the levels of 25(OH)D were compared between women who subsequently suffered spontaneous abortions (n=59) and the rest of the population, corrected for select covariates.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and residing in the municipality of Odense during 2010-2012

Exclusion Criteria:

* Not residing in Odense, leaving the municipality

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Odense Child Cohort Study (OCC) is a population-based cohort study, comprising pregnant women recruited between January 1st 2010 and December 31st 2012. All women who were pregnant in the municipality of Odense during this time were eligible for participation, and 6,707 women were approached directly with recruitment material.
  The study complied with the Helsinki declaration and was approved by the Regional Scientific Ethical Committee for Southern Denmark, no. S-20090130. All participants gave informed consent. From a population base of 6,70 pregnant women, 2,874 (42.9%) enrolled in the OCC up to December 31st, 2012. The children will be followed until 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 2874 (Actual)
Dates: Start 2010-01; Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Spontaneous Abortion | Outcome is assessed in gestational weeks 5+0 to 22+0.
  Occurrence of spontaneous abortion, as diagnosed by transvaginal ultrasound in medical files. The time from inclusion in cohort to occurrance of spontaneous abortion was on average 13 days.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik T Christesen, MD, PhD, Principal Investigator — Project leader
Locations (1):
- HCA Research, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Galthen-Sorensen M, Andersen LB, Sperling L, Christesen HT. Maternal 25-hydroxyvitamin D level and fetal bone growth assessed by ultrasound: a systematic review. Ultrasound Obstet Gynecol. 2014 Dec;44(6):633-40. doi: 10.1002/uog.13431. PMID 24891235
- [Background] Christesen HT, Elvander C, Lamont RF, Jorgensen JS. The impact of vitamin D in pregnancy on extraskeletal health in children: a systematic review. Acta Obstet Gynecol Scand. 2012 Dec;91(12):1368-80. doi: 10.1111/aogs.12006. PMID 23210535
- [Background] Christesen HT, Falkenberg T, Lamont RF, Jorgensen JS. The impact of vitamin D on pregnancy: a systematic review. Acta Obstet Gynecol Scand. 2012 Dec;91(12):1357-67. doi: 10.1111/aogs.12000. Epub 2012 Oct 17. PMID 22974137
- [Result] Christesen HT, Andersen LB. Reply to: 'vitamin D deficiency during pregnancy: confronting the issues'. Clin Endocrinol (Oxf). 2014 Jul;81(1):155-6. doi: 10.1111/cen.12328. Epub 2013 Oct 15. No abstract available. PMID 24102268
- [Result] Andersen LB, Abrahamsen B, Dalgard C, Kyhl HB, Beck-Nielsen SS, Frost-Nielsen M, Jorgensen JS, Barington T, Christesen HT. Parity and tanned white skin as novel predictors of vitamin D status in early pregnancy: a population-based cohort study. Clin Endocrinol (Oxf). 2013 Sep;79(3):333-41. doi: 10.1111/cen.12147. Epub 2013 Jul 2. PMID 23305099
- [Derived] Andersen LB, Jorgensen JS, Jensen TK, Dalgard C, Barington T, Nielsen J, Beck-Nielsen SS, Husby S, Abrahamsen B, Lamont RF, Christesen HT. Vitamin D insufficiency is associated with increased risk of first-trimester miscarriage in the Odense Child Cohort. Am J Clin Nutr. 2015 Sep;102(3):633-8. doi: 10.3945/ajcn.114.103655. Epub 2015 Jul 15. PMID 26178723